CLINICAL TRIAL: NCT07337551
Title: Gossypol Acetate Combined With Bevacizumab and FOLFIRI as Second-Line Therapy for Metastatic Colorectal Cancer With TP53 Mutation and LRPPRC Positivity: A Single-Center, Single-Arm Clinical Study
Brief Title: Gossypol Acetate + FOLFIRI + Bev in mCRC With TP53-Mutant and LRPPRC Positive
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guiying Wang (Other)
Responsible Party: Sponsor-Investigator, Guiying Wang, Chief Physician, Professor, The Second Hospital of Hebei Medical University
Organization: The Second Hospital of Hebei Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-R689
Record Dates: First submitted 2025-08-27; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Patients With Metastatic Colorectal Cancer Who Were TP53-mutant and LRPPRC-positive and Had Previously Failed Prior First-line Treatment
Keywords: TP53 mutant; LRPPRC positive; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- GAA+FOLFIRI + Bev (Experimental)
  Interventions: Drug: Gossypol acetate Combined with Bevacizumab and FOLFIRI

INTERVENTIONS:
Drug: Gossypol acetate Combined with Bevacizumab and FOLFIRI — Gossypol Acetate Oral 20mg/day

SUMMARY:
This study is a single-center, single-arm clinical trial involving patients with TP53-mutated and LRPPRC-positive metastatic colorectal cancer. It aims to evaluate the efficacy and safety of gossypol acetate tablets combined with bevacizumab and the FOLFIRI regimen as a second-line treatment. The study is based on a key scientific finding: LRPPRC is a critical protein mediating chemotherapy resistance induced by TP53 mutation, and gossypol acetate-an existing drug-can specifically degrade LRPPRC. Preclinical studies have demonstrated its potential to effectively reverse drug resistance.

Patients who have experienced failure of first-line oxaliplatin-based therapy are planned to be enrolled. All eligible subjects will receive the same combined treatment regimen until disease progression or unacceptable toxicity occurs. The primary endpoint is objective response rate (ORR), and secondary endpoints include progression-free survival (PFS), overall survival (OS), and safety. Throughout the treatment period, patients will undergo regular tumor imaging evaluations and safety monitoring. Statistical analyses will be performed using both the full analysis set and the per-protocol set.

This study strictly adheres to ethical standards and aims to explore a new potential treatment strategy for this specific refractory patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged ≥18 years.
2. Histopathologically or cytologically confirmed adenocarcinoma of the colon or rectum.
3. Radiologically confirmed unresectable metastatic disease.
4. At least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Prior first-line treatment with an oxaliplatin-based regimen.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
7. Life expectancy ≥3 months.
8. Adequate bone marrow function: absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count (PLT) ≥100×10⁹/L, hemoglobin (Hb) ≥90 g/L, and white blood cell count (WBC) ≥3.0×10⁹/L.
9. Adequate liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) ≤2.5 × the upper limit of normal (ULN), or ≤5×ULN in the presence of liver metastases; total bilirubin ≤1.5×ULN.
10. Adequate renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance ≥60 mL/min (calculated using the Cockcroft-Gault formula), and urine protein <2+.
11. Normal coagulation function: international normalized ratio (INR) ≤1.5.
12. Ability to understand the study requirements; voluntary provision of written informed consent by the patient and/or legal representative.

Exclusion Criteria:

1. Patients with a history of other malignant tumors within the past 5 years (except cured carcinoma *in situ* or basal cell carcinoma of the skin).
2. Patients previously subjected to irinotecan or irinotecan liposome-based chemotherapy.
3. Presence of massive pleural effusion or ascites requiring therapeutic intervention.
4. Active, uncontrolled bacterial, viral, or fungal infection requiring systemic treatment, defined as persistent signs/symptoms related to the infection without improvement despite appropriate antibiotic, antiviral, and/or other therapy.
5. Known active HIV infection (i.e., positive for HIV-1/2 antibodies); untreated active HBV infection (defined as positive for HBsAg or HBcAg with detectable HBV-DNA copies exceeding the upper limit of normal [ULN] at the local laboratory) and active HCV infection (positive for HCV antibody with an HCV-RNA level above the ULN).
6. Concurrent uncontrolled systemic diseases, including cardiovascular disorders such as unstable angina, myocardial infarction, congestive heart failure, severe unstable ventricular arrhythmias, or a history of severe pericardial disease; uncontrolled hypertension (defined as systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg after standardized antihypertensive therapy) or a history of hypertensive crisis or hypertensive encephalopathy; uncontrolled diabetes mellitus, etc.
7. Presence of severe gastrointestinal diseases (including active bleeding, obstruction greater than Grade 1, diarrhea greater than Grade 1, or gastrointestinal perforation).
8. History of laparotomy, thoracotomy, or intestinal resection within 28 days prior to enrollment.
9. Presence of interstitial lung disease or pulmonary fibrosis.
10. Known allergy or intolerance to the investigational drug(s) or their excipients.
11. History of pulmonary hemorrhage/hemoptysis ≥ Grade 2 (defined as at least 2.5 mL of bright red blood) within one month prior to enrollment.
12. History of arterial thromboembolism, severe hemorrhage (excluding bleeding due to surgery), or current predisposition to embolism or severe hemorrhage within 6 months prior to enrollment.
13. Presence of central nervous system metastases.
14. Serum albumin level ≤ 3 g/dL.
15. Concomitant use of strong inhibitors or inducers of CYP3A4, CYP2C8, or UGT1A1.
16. Pregnant or lactating women, as well as patients of childbearing potential who refuse to adopt adequate contraceptive measures during the trial.
17. Participation in another clinical trial within 30 days prior to the first dose of the investigational drug.
18. Allergy to bevacizumab, irinotecan, fluorouracil, calcium folinate, or compound gossypol acetate tablets.
19. Patients deemed by the investigator to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | up to 16 months
  Objective Response Rate (ORR)

SECONDARY OUTCOMES:
Secondary Endpoints | up to 16 months
  Progression-Free Survival (PFS)
Secondary Endpoints | up to 16 months
  Clinical Benefit Rate (CBR)
Secondary Endpoints | up to 16 months
  Duration of Response (DoR)
Secondary Endpoints | up to 16 months
  Time to Response (TTR)
Secondary Endpoints | up to 16 months
  Overall Survival (OS)
Secondary Endpoints | up to 16 months
  Adverse Events (AE)

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2026-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT07337551/Prot_000.pdf
  • Informed Consent Form (2026-01-04): https://cdn.clinicaltrials.gov/large-docs/51/NCT07337551/ICF_001.pdf